CLINICAL TRIAL: NCT01210391
Title: Assessment of Growth of Infants Fed a 100% Whey Extensively Hydrolyzed Formula.
Brief Title: Growth of Infants Fed an Extensively Hydrolyzed Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 09.43.PED
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Growth
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New hydrolyzed infant formula (Experimental): New, extensively hydrolyzed infant formula
  Interventions: Other: Extensively hydrolyzed whey infant formula
- Commercially available infant formula (Active Comparator): Commercially available, extensively hydrolyzed infant formula.
  Interventions: Other: Extensively hydrolyzed casein infant formula

INTERVENTIONS:
Other: Extensively hydrolyzed whey infant formula — New hydrolyzed infant formula.
  Other Names: Baby Formula
  Arms: New hydrolyzed infant formula
Other: Extensively hydrolyzed casein infant formula — Commercially available infant formula.
  Other Names: Baby Formula
  Arms: Commercially available infant formula

SUMMARY:
The primary objective of the clinical trial is to compare growth in infants (expressed as weight gain in g/day) consuming a new extensively hydrolyzed formula (EHF) to infants consuming a commercially available EHF.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn singleton infant
* Full-term (>= 37 weeks gestation)
* Birth weight between >= 2500 and < =4500 g
* 14 ± 3 days of age on enrollment
* Infant's mother has elected not to breastfeed
* baby has been exclusively formula fed a minimum of 3 days prior to enrollment
* Study explained and written information provided with Parent/Caregiver
* Informed consent signed (parent/legal representative)

Exclusion Criteria:

* Congenital illness or malformation affecting infant feeding and/or growth
* Suspected or known allergy to cow's milk protein
* Significant pre-natal and/or post-natal disease
* Any readmission to hospital (except for hyperbilirubinemia) prior to enrollment
* Infant has received oral or IV antibiotic therapy in the 10 days prior to enrollment
* Infant receiving prescription medication (with exception of topical antibiotics and/or treatment for thrush) or frequent use of over the counter medications except vitamin and mineral supplements
* Infant has received probiotics in the seven days prior to enrollment
* Infant currently participating in another clinical study
* Infant's family who in the Investigator's assessment cannot be expected to comply with the protocol

Ages: 11 Days to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Weight Gain | 4 Months
  Mean weight gain (g/day) from enrollment to 4 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Sorensen, MD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (20):
- United States (20):
  - Colorado Springs Health Partners, Colorado Springs, Colorado
  - Pedia Research, Newburgh, Indiana
  - Pedia Research, Owensboro, Kentucky
  - ARK-LA-Tex Pediatric Research, Bossier City, Louisiana
  - The Clinical Trials Center, New Orleans, Louisiana
  - Clinical Research of Nevada, Las Vegas, Nevada
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Square-1 Clinical Research, Erie, Pennsylvania
  - Alpha Clinical Research, Clarksville, Tennessee
  - Jackson Clinic, Jackson, Tennessee
  - Scott & White Wells Branch Clinic, Austin, Texas
  - Scott & White Killeen Clinic, Killeen, Texas
  - DCOL Center for Research, Longview, Texas
  - Southwest Children's Research Associates, San Antonio, Texas
  - Scott & White Temple, Temple, Texas
  - Tanner Clinic, Layton, Utah
  - Clinical Research Partners, Richmond, Virginia
  - Wenatchee Valley Medical Center, Wenatchee, Washington